CLINICAL TRIAL: NCT03974282
Title: Brain Function and Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20015724; UL1TR002649 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Behavior, Social; Psychology, Social; Social Interaction; Interpersonal Relations
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low psychopathy distribution (Other): Participants who score at the low end of the psychopathy distribution
  Interventions: Behavioral: Psychological task
- High psychopathy distribution (Other): Participants who score at the high end of the psychopathy distribution
  Interventions: Behavioral: Psychological task

INTERVENTIONS:
Behavioral: Psychological task — Participants will complete a psychological task that evokes antisocially- and prosocially-motivated empathic responding

SUMMARY:
This study is about how brain function and structure is different between two universities. Participant in this project will contribute to a better understanding of how universities affect the brain.

DETAILED DESCRIPTION:
Some study details are purposely omitted at this time to preserve scientific integrity. Now that the study is completed, full details are included below.

The true purpose of this study was to investigate the psychometric properties of the two computer tasks that participants completed. Specifically, researchers wanted to know if they would be able to accurately measure motivated empathy. To better understand this, participants were asked to rate images of people expressing pain and were told that these were either students from their university or students from a different university. This was not the case. The faces shown were random images produced for a research study.

Researchers also wanted to know if they could accurately measure moral decision making and how those judgments relate to aggression. To examine this, participants were asked whether various scenarios were immoral and then asked about aggressive tendencies.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students aged 18 - 35 years of age
* No current or regular use of prescribed or illicit psychoactive drugs
* Free of major health problems (e.g., diabetes, HIV, Parkinson's disease)
* Free of a neurological or psychiatric disorders
* No current drug abuse (e.g., recreational drug use, average alcohol intake in excess of 4 drinks per day).
* Right hand dominant
* Free of claustrophobia
* Free of pregnancy or suspected pregnancy
* Absent MRI risk factors (e.g., implanted medical device, body mass index > 35, braces)
* Free of medical conditions that render individuals with overly sensitive hearing
* No colorblindness

Exclusion Criteria:

• Not meeting the inclusion criteria listed above.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chester, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Psychopathy Distribution | High Psychopathy Distribution
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Psychopathy Distribution | High Psychopathy Distribution | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.24 (2.75) | 20.59 (2.12) | 20.41 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 5 | 8
  Race: Black or African-American | 5 | 1 | 6
  Race: Pacific Islander | 1 | 0 | 1
  Race: White - Hispanic | 3 | 1 | 4
  Race: Missing Data | 1 | 1 | 2
  Race: Multiracial | 1 | 0 | 1
  Race: Other Race | 2 | 0 | 2
  Race: White - Non-Hispanic | 2 | 10 | 12
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Prefrontal Cortex Brain Activity Assessed by fMRI
Description: Blood-Oxygen-Level-Dependent signal change in the cognitive empathy brain network will be assessed using functional MRI
Time Frame: Baseline to 3 hours
Measure: Mean (Standard Deviation); unit: Percent BOLD Signal Change
Arm/Group | Low Psychopathy Distribution | High Psychopathy Distribution
Number analyzed (Participants) | 18 | 18
Percent BOLD Signal Change | -0.002 (0.163) | 0.015 (0.105)

2. Primary Outcome: Change in Accuracy of Empathic Pain Judgments
Description: Difference in pain judgment scores rated from 1 (low) to 4 (high) between antisocial vs prosocial empathy trials
Time Frame: Baseline to 3 hours
Measure: Mean (Standard Deviation); unit: difference in pain scores
Arm/Group | Low Psychopathy Distribution | High Psychopathy Distribution
Number analyzed (Participants) | 18 | 18
difference in pain scores | .49 (.14) | .39 (.14)

ADVERSE EVENTS:
Time Frame: 3 hours
Groups:
- All Participants: Participants who score at the low or high end of the psychopathy distribution
  Because all participants received the same intervention, adverse events were not recorded separately by arm.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT03974282/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03974282/ICF_000.pdf